CLINICAL TRIAL: NCT02315794
Title: Aesthetic Outcomes of Single Tooth Implant-supported Restorations Using Metal Ceramic Restorations With Either Zirconia or Titanium Abutments: A Randomized Controlled Clinical Study
Brief Title: Aesthetic Outcomes of Single Tooth Implant Using Metal Ceramic Restorations With Either Zirconia or Titanium Abutments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Firenze and Siena, Napoli, Italy (Other)
Responsible Party: Principal Investigator, nicola baldini, oral surgeon, University of Firenze and Siena, Napoli, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aostirct
Record Dates: First submitted 2014-12-06; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Thick Gingival Margin to Tooth Restoration
Keywords: aesthetic outcome; titanium abutment; zirconia abutment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPI®ART (Experimental): in test group after a three month healing period a zirconia abutment was connected to the implant to realize the prosthetic restoration
  Interventions: Device: SPI®ART
- SPI®EASY (Active Comparator): in control group a three month healing period a titanium abutment was connected to the implant for the prosthetic restoration
  Interventions: Device: SPI®EASY

INTERVENTIONS:
Device: SPI®ART — implant prothetic restoration using a yttrium oxide stabilized zirconia abutment
  Arms: SPI®ART
Device: SPI®EASY — implant prosthetic restoration using a commercially pure titanium grade 4 abutment
  Arms: SPI®EASY

SUMMARY:
Different studies have proposed the use of zirconia abutments to improve the aesthetic outcomes in the anterior sextant, however the results have been inconclusive. A tendency towards a better aesthetic result with the use of zirconia instead of titanium abutments was observed, although more technical complications were also recorded.The use of zirconia abutments in the anterior maxillary region showed a tendency towards better matching, although differences were not significant. In addition, with these abutments more technical complications were observed, what increased the cost and time. More studies with larger samples and longer observations periods are needed to recommend the use of zirconia abutments for this clinical situation

DETAILED DESCRIPTION:
The purpose of the present study was to evaluate the clinical and aesthetic outcomes of single tooth implant restorations, where different abutment materials were used (zirconia vs titanium) associated with metal-ceramic crowns. The evaluation was carried out by means of an aesthetic composite index combined with patient evaluation

ELIGIBILITY:
Inclusion Criteria:

* mono-edentulism condition in the aesthetic zone
* minimum of 2 mm of keratinized gingiva

Exclusion Criteria:

* systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change from baseline in the anatomic form and surface characteristics of the peri implant mucosa | one month and one year after the placement of the definitive crowns
  the following parameters were assessed by means of standardized photographs: contour of the labial surface of the mucosa and its colour; when compared to the adjacent teeth , penalty points were assigned ( 0 = excellent; 1 or 2 = satisfactory; 3 or 4 = moderate; 5 ore more, poor).

SECONDARY OUTCOMES:
change from baseline in crestal bone levels | one month and one year after placing the definitive crown
  in standardized intraoral radiographs the the following measurements were carried out : vertical distance from implant shoulder to the most coronal bone in contact with the implant at mesial and distal site; horizontal distance from the implant shoulder to the adjacent teeth at mesial and distal sites; vertical distance ( parallel to the implant long axis) from the contact point to the bone crest at mesial and distal sides
change from baseline in interdental soft tissue position | one month and one year after the placement of the definitive crowns
  position of interdental papilla measured by means of Papilla Index ( Jemt, 1997)
change from baseline in thickness of the peri implant mucosa | one month and one year after the placement of the definitive crowns
  the thickness was measured by placing a calibrated endodontic file 2mm apical to the mucosal margin

CONTACTS AND LOCATIONS:
Overall Officials: nicola baldini, oral surgeon, Principal Investigator — tuscal school of dental medicine
Locations (2):
- Italy (2):
  - Siena University, Department of Periodontology, Policlinico Le Scotte Siena., Siena, Siena
  - Tuscan School of Dentistry, Siena, Siena

REFERENCES:
- [Background] Meijer HJ, Stellingsma K, Meijndert L, Raghoebar GM. A new index for rating aesthetics of implant-supported single crowns and adjacent soft tissues--the Implant Crown Aesthetic Index. Clin Oral Implants Res. 2005 Dec;16(6):645-9. doi: 10.1111/j.1600-0501.2005.01128.x. PMID 16307570
- [Derived] Ferrantino L, Carrillo de Albornoz A, Sanz M. Five-year outcomes of a randomized controlled clinical trial comparing single-tooth implant-supported restoration with either zirconia or titanium abutments. J Clin Periodontol. 2023 Jun;50(6):744-754. doi: 10.1111/jcpe.13787. Epub 2023 Feb 28. PMID 36748305